CLINICAL TRIAL: NCT03584542
Title: Impact of Regulatory Framework Change for Zolpidem Prescriptions (Secure Prescription) on Consumption and Misuse of Sedatives Drugs.
Brief Title: ZOlpidem and the stRengthening of pRescription regulatiOn
Acronym: ZORRO
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0381
Record Dates: First submitted 2018-06-12; First posted 2018-07-12 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Substance Use Disorders
Keywords: Zolpidem; hypnotics and sedatives; Drug and narcotic control; Drug prescription; Substance-related Disorders; Health Impact Assessment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients in general practitioners' offices: No interventional study. Only one questionnaire will be done
  Interventions: Other: No interventional study
- Patients of specialized centers for drug addict patients: No interventional study Only one questionnaire will be done
  Interventions: Other: No interventional study
- General practitioners: No interventional study Only one questionnaire will be done
  Interventions: Other: No interventional study

INTERVENTIONS:
Other: No interventional study — No Interventional study - Only one questionnaire will be done for patients and for general practitioners

SUMMARY:
For several years, the French Addictovigilance Network (FAN) highlights potential problematic consumptions with zolpidem. To prevent abuse and misuse of zolpidem, the French Health Products Agency has changed the regulatory framework of zolpidem prescription. Thus, since the 10th of April 2017 zolpidem prescriptions have to be secured (particular support, dosage written out). The investigators hypothesized that this change will affect zolpidem consumption but also the consumption of all sedative drugs. In order to assess the incidence of the regulatory change for zolpidem prescription the investigators conduct a two part study: an epidemiological study with French National Health Insurance Fund for Employees database and an observational study with general practitioners and zolpidem consumers.

DETAILED DESCRIPTION:
Several aspects of the incidence will be assessed (number of zolpidem consumers, change in consumption profile, and consumption of other sedative drugs) before and after the regulatory framework change.

The epidemiological study will enable us to respond to all these aspects and it will be completed by the observational study with practitioners and patients that have been affected by the regulatory framework change.

General practitioners will be interviewed by phone about their perception of the regulatory framework change, their attitudes towards their patients with zolpidem prescription and the drugs they used if they had changed the patients prescription.

All consumers included in the study will have to fulfill a self-questionnaire about their perception of the regulatory framework change, their attitudes towards their consumption of zolpidem (stop, diminution, replacement) and their favorite replacement drug.

The impact of regulatory prescription change of zolpidem will have a pleiotropic impact which can't be evaluated on a single criterion. It must be considered in a global, multifocal manner. This is why several criteria will be used to assess several incidence and several populations.

These different approaches will enable us to respond to three questions

* What is the impact on the number of consumers? Prevalence and incidence of zolpidem consumers over several periods (before and after the regulatory prescription change) will be evaluated from French National Health Insurance Fund for Employees database.
* What is the impact on consumption patterns of zolpidem? The investigators will assess different patterns of zolpidem consumption (i) occasional use versus chronic use will be assessed from French National Health Insurance Fund for Employees database and from consumers of general medicine and specialized centers for drug addict patients (ii) problematic use (consumption not in accordance with summary of product characteristics according to at least one of these parameters: duration of consumption, dosage, manner in which zolpidem is obtained, route of administration, or seeking psychoactive effects different from hypnotic effect) versus no problematic use will be assessed from French National Health Insurance Fund for Employees database and from consumers of general medicine and specialized centers for drug addict patients.
* What is the impact on consumption of other sedatives drugs? The investigators will look for reports of zolpidem prescriptions on other drugs and if reports are maintained from French National Health Insurance Fund for Employees database, general practitioners will be interviewed about change in their prescriptions and their preferred drug for replacement, and consumers of general medicine and specialized centers for drug addict patients will be asked about their attitudes towards their consumption of zolpidem (stop, diminution, replacement) and their favorite replacement drug.

ELIGIBILITY:
Inclusion Criteria:

Epidemiological study: all the patients of the database between January 2016 and December 2018 will be selected.

Observational study with general practitioners:

* General practitioners drawn by the sampling methodology or general practitioners that are habitual partners of the investigator service.
* General practitioners located in liberal cabinet when the change in regulatory framework has been applied.
* General practitioners who accept the interview.

Observational study with zolpidem consumers:

* Being a patient from one of the general practitioners participating in the study or going in one of the specialized centers for drug addict patients participating in the study.
* Having a problematic consumption of zolpidem when the regulatory framework change was applied according to the general practitioner or to the specialized centre staff.
* Giving consent oral to participate.

Exclusion Criteria:

Epidemiological study: none

Observational study with general practitioners:

- General practitioners who not respond to the phone call after several attempts.

Observational study with zolpidem consumers:

* being under 18 years of age
* being an adult protected
* having difficulties to understand, read or write French language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the epidemiological study: all the patients of the database between January 2016 and December 2018 will be selected.
  For the observational study with general practitioners: 100. For the observational study with zolpidem consumers from general medicine and specialized centers for drug addict patients: 400 (200 from general medicine and 200 from specialized centres).
Sampling Method: Non-Probability Sample
Enrollment: 449 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of zolpidem consumers and substance use disorders with zolpidem (according to the number of DSM 5 criteria) before and after the regulatory prescription change | Day 1
  The impact of regulatory prescription change of zolpidem will have a pleiotropic impact which can't be evaluated on a single criterion. It must be considered in a global, multifocal manner. This is why several criteria will be used to assess several incidence and several populations.
  These different approaches will enable us to respond to three questions
  * What is the impact on the number of consumers?
  * What is the impact on consumption patterns of zolpidem?
  * What is the impact on consumtion of other sedative drugs? Cf "detailed desciption" paragraph

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

REFERENCES:
- [Derived] Istvan M, Rousselet M, Laforgue EJ, Guerlais M, Gerardin M, Jolliet P, Feuillet F, Victorri-Vigneau C. Did the pattern of use of zolpidem change since the enforcement of a new prescription rule? A latent class analysis using the French health insurance database. Expert Opin Drug Saf. 2022 Sep;21(9):1225-1234. doi: 10.1080/14740338.2022.2047930. Epub 2022 Mar 8. PMID 35255750
- [Derived] Gerardin M, Rousselet M, Caillet P, Grall-Bronnec M, Loue P, Jolliet P, Victorri-Vigneau C. French national health insurance database analysis and field study focusing on the impact of secure prescription pads on zolpidem consumption and sedative drug misuse: ZORRO study protocol. BMJ Open. 2019 Jun 28;9(6):e027443. doi: 10.1136/bmjopen-2018-027443. PMID 31256026